CLINICAL TRIAL: NCT05342610
Title: Effect of Reiki Application on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Didem Lafci, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUnivers
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Menopausal Symptom
Keywords: Nursing; integrative practice; menopausal symptoms; reiki
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (distant reiki) group (Experimental): Reiki (complementary and integrative medicine method) was applied individually to the experimental group for 30 minutes three times a week for four weeks. Data collection forms was applied 3 times in total, before the intervention, in the fourth and the eighth week.
  Interventions: Other: Distant reiki
- Control group (No Intervention): No intervention was made to women in the control group. However, data collection forms was applied 3 times in total, before the intervention, in the fourth and the eighth week.

INTERVENTIONS:
Other: Distant reiki — Reiki; It is the transfer of energy to other people by the hands of the person who receives the theoretical training and attunement (initiation) from the reiki master, close or distant. When the hands are brought closer to the body in suitable positions or when the reiki practitioner visualizes the person in his/her thoughts, the energy flow starts spontaneously and the transferred energy is shaped according to the needs of the reiki recipient. The biggest advantage of Reiki; It is an easy and cost-effective method to ensure that the individual restores the balance between body, mind and spirit, has no side effects, has no negative effects on behavior and attitudes.
  Other Names: Reiki
  Arms: Experimental (distant reiki) group

SUMMARY:
In this randomized controlled study, it was aimed to determine the effect of distant reiki on menopausal symptoms. Two different hypothesis teams have been established for the study.

These; H0: There is no significant difference between the menopause rating scores of the women in the study group in which distant reiki was applied and the control group without distant reiki.

H1: There is a significant difference between the menopause rating scores of the women in the study group in which distant reiki was applied and the control group without distant reiki.

DETAILED DESCRIPTION:
Parallel to the increase in life expectancy by years, the population of women living in the post-menopausal period is also increasing. In order to have a healthy menopause, which is an important part of women's life, it is thought that the distant reiki without health risks by women may be effective in reducing the symptoms of menopause experienced by women. In line with this information, it was aimed to determine the effect of distant reiki on menopausal symptoms. The study was carried out with menopausal women between the ages of 40-55 in Adana province in Turkey. Therefore, in the study, 48 women in the menopausal period between the ages of 40-55 was randomly assigned to reiki and control groups. Distant reiki application for 30 minutes three times a week for four weeks was applied individually to the study group. No intervention was made to the control group for a period of four weeks. The primary expected outcome of the research is the effect of distant reiki on menopausal symptoms of menopausal women. Results was applied three times in total, before the study and control application, 4 weeks and 8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in research,
* Can read and write in Turkish,
* Open to communication,
* Those who are between the ages of 40-55 and do not experience menstruation for at least one year,
* Experiencing at least one or more of the menopausal symptoms,
* Not applying regular reiki,
* Those who have not surgically entered menopause,
* Women without psychiatric problems

Exclusion Criteria:

* Who do not agree to participate in the research,
* Can't read and write Turkish,
* Communication is not possible,
* Those who are younger than 40, older than 55, have experienced menstruation for at least one year,
* Do not experience the symptoms of menopause,
* Using medication for the treatment of menopausal symptoms,
* Chronic illness,
* Regular reiki is applied,
* Surgically in menopause,
* Women with psychiatric problems

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 40-55 who are in menopause
Enrollment: 48 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Menopause symptoms evaluated using the Menopause Rating Scale | Change from before intervention, 4th and 8th week of intervention
  It was developed in German by Schneider et al. In 1992 to measure the severity of menopausal symptoms and was adapted to English in 1996. MRT was adapted to Turkish by Gürkan in our country in 2005. There are "0 = None", "1 = Mild", "2 = Moderate", "3 = Severe" and "4 = Very severe" options for each item in the Likert-type scale consisting of 11 items including menopausal complaints. The total score of the scale is calculated based on the scores given for each item. The lowest score that can be obtained from the scale is 0, the highest score is 44.

CONTACTS AND LOCATIONS:
Locations (1):
- Diğdem LAFCI, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No